CLINICAL TRIAL: NCT04655391
Title: A Pilot/Phase 1b Study of Glasdegib-Based Treatment Combinations in Adult Patients With Relapsed AML Post Allogeneic Hematopoietic Cell Transplantation
Brief Title: Glasdegib-Based Treatment Combinations for the Treatment of Patients With Relapsed Acute Myeloid Leukemia Who Have Undergone Hematopoietic Cell Transplantation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug availability
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20456; NCI-2020-10595 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20456 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — bosutinib; Decitabine; Injections; 2-Propanol; methanesulfonic acid; enasidenib; gilteritinib; glasdegib; ivosidenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Chapter 1 (glasdegib, decitabine, venetoclax) (Experimental): MOLECULAR DIAGNOSIS SEGMENT: Patients receive glasdegib PO QD for at least 14 days until their AML TAC recommendation is made and they are either consented to a treatment arm in the Treatment Segment or go off study.
  TREATMENT SEGMENT: Patients receive glasdegib PO QD on days 1-28,decitabine IV over 1 hour on days 1-5, and venetoclax PO QD on days 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Drug: Glasdegib Maleate; Drug: Venetoclax
- Chapter 2 (glasdegib, gilteritinib) (Experimental): MOLECULAR DIAGNOSIS SEGMENT: Patients receive glasdegib PO QD for at least 14 days until their AML TAC recommendation is made and they are either consented to a treatment arm in the Treatment Segment or go off study.
  TREATMENT SEGMENT: Patients receive glasdegib PO QD and gilteritinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gilteritinib Fumarate; Drug: Glasdegib Maleate
- Chapter 3 (glasdegib, bosutinib) (Experimental): MOLECULAR DIAGNOSIS SEGMENT: Patients receive glasdegib PO QD for at least 14 days until their AML TAC recommendation is made and they are either consented to a treatment arm in the Treatment Segment or go off study.
  TREATMENT SEGMENT: Patients receive glasdegib PO QD and bosutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosutinib Monohydrate; Drug: Glasdegib Maleate
- Chapter 4 (glasdegib, ivosidenib) (Experimental): MOLECULAR DIAGNOSIS SEGMENT: Patients receive glasdegib PO QD for at least 14 days until their AML TAC recommendation is made and they are either consented to a treatment arm in the Treatment Segment or go off study.
  TREATMENT SEGMENT: Patients receive glasdegib PO QD and ivosidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Glasdegib Maleate; Drug: Ivosidenib
- Chapter 5 (glasdegib, enasidenib) (Experimental): MOLECULAR DIAGNOSIS SEGMENT: Patients receive glasdegib PO QD for at least 14 days until their AML TAC recommendation is made and they are either consented to a treatment arm in the Treatment Segment or go off study.
  TREATMENT SEGMENT: Patients receive glasdegib PO QD and enasidenib PO QD on days 1-28 .Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enasidenib Mesylate; Drug: Glasdegib Maleate

INTERVENTIONS:
Drug: Bosutinib Monohydrate — Given PO
  Other Names: 3-Quinolinecarbonitrile, 4-((2,4-Dichloro-5-methoxyphenyl)amino)-6-methoxy-7-(3-(4-methyl-1-piperazinyl)propoxy)-, Hydrate (1:1); Bosulif; SKI-606 Monohydrate
  Arms: Chapter 3 (glasdegib, bosutinib)
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: Chapter 1 (glasdegib, decitabine, venetoclax)
Drug: Enasidenib Mesylate — Given IV
  Other Names: 2-Methyl-1-[(4-[6-(trifluoromethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyridin-4-yl]amino}-1,3,5-triazin-2-yl)amino]propan-2-ol Methanesulfonate; 2-Propanol, 2-Methyl-1-((4-(6-(trifluoromethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triazin-2-yl)amino)-, Methanesulfonate (1:1); AG-221 Mesylate; CC-90007; Enasidenib Methanesulfonate; Idhifa
  Arms: Chapter 5 (glasdegib, enasidenib)
Drug: Gilteritinib Fumarate — Given PO
  Other Names: ASP-2215 Hemifumarate; ASP2215 Hemifumarate; Gilteritinib Hemifumarate; Xospata
  Arms: Chapter 2 (glasdegib, gilteritinib)
Drug: Glasdegib Maleate — Given PO
  Other Names: Daurismo; PF 04449913 Maleate
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo
  Arms: Chapter 4 (glasdegib, ivosidenib)
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
  Arms: Chapter 1 (glasdegib, decitabine, venetoclax)

SUMMARY:
This phase Ib trial evaluates the best dose and effect of glasdegib in combination with venetoclax and decitabine, or gilteritinib, bosutinib, ivosidenib, or enasidenib in treating patients with acute myeloid leukemia that has come back (relapsed) after stem cell transplantation. Chemotherapy drugs, such as venetoclax and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Glasdegib, bosutinib, ivosidenib, and enasidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Glasdegib inhibits the Sonic the Hedgehog gene. Venetoclax inhibits BCL-2 gene. Bosutinib is a tyrosine kinase inhibitor that inhibits BCR-ABL gene fusion. Ivosidenib inhibits isocitrate dehydrogenase-1 gene or IDH-1. Enasidenib inhibits isocitrate dehydrogenase-2 gene or IDH-2. This study involves an individualized approach that may allow doctors and researchers to more accurately predict which treatment plan works best for patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate study feasibility through:

Ia. The ability to obtain a molecular diagnosis within 10 calendar days from study enrollment in at least 90% of participants. (Molecular Diagnosis Segment) Ib. The ability to make a treatment arm assignment within 14 calendar days from study enrollment in at least 90% of participants. (Molecular Diagnosis Segment) II. Assess the safety and tolerability of the drug combination by evaluation of toxicities including: type, frequency, severity, attribution, and duration of the toxicity. (Treatment Segment)

SECONDARY OBJECTIVES:

I. Determine the proportion of participants with successful sequencing by City of Hope (COH) Pathology among those with less than 10% blasts in the marrow aspirate. (Molecular Diagnosis Segment) II. Determine the proportion of participants with successful treatment arm registration based on Treatment Assignment Committee (TAC) assignment. (Molecular Diagnosis Segment) III. Assess the safety of monotherapy glasdegib by evaluation of toxicities including, type, frequency, severity and attribution. (Molecular Diagnosis Segment) IV. Obtain preliminary estimates of remission (complete response [CR] + CR with incomplete blood count recovery [CRi]) rate and duration of remission. (Treatment Segment)

EXPLORATORY OBJECTIVE:

I. Measure and characterize the leukemia stem cell (LSC) burden. (Treatment Segment)

OUTLINE: This is a dose escalation study of glasdegib maleate (glasdegib) followed by a dose-expansion study.

MOLECULAR DIAGNOSIS SEGMENT: Patients receive glasdegib orally (PO) once daily (QD) for at least 14 days until their acute myeloid leukemia (AML) TAC recommendation is made and they are either consented to a treatment arm in the Treatment Segment or go off study.

TREATMENT SEGMENT: Patients are assigned to 1 of 5 arms.

CHAPTER 1: Patients receive glasdegib PO QD on days 1-28, decitabine intravenously (IV) over 1 hour on days 1-5, and venetoclax PO QD on days 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

CHAPTER 2: Patients receive glasdegib PO QD and gilteritinib fumarate (gilteritinib) PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

CHAPTER 3: Patients receive glasdegib PO QD and bosutinib monohydrate (bosutinib) PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

CHAPTER 4: Patients receive glasdegib PO QD and ivosidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

CHAPTER 5: Patients receive glasdegib PO QD and enasidenib mesylate (enasidenib) PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* MOLECULAR DIAGNOSIS SEGMENT: Documented informed consent of the participant and/or legally authorized representative
* MOLECULAR DIAGNOSIS SEGMENT: Age: >= 18 years on the day of signing informed consent
* MOLECULAR DIAGNOSIS SEGMENT: Eastern Cooperative Oncology Group (ECOG) =< 2
* MOLECULAR DIAGNOSIS SEGMENT: Patients with histologically confirmed acute myeloid leukemia (AML), according to World Health Organization (WHO) criteria, with relapsed disease after allogeneic hematopoietic cell transplantation (alloHCT)

  * Patients with non-central nervous system (CNS) extramedullary disease may be included if they also have marrow disease
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
* MOLECULAR DIAGNOSIS SEGMENT: Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 of prior anti-cancer therapy
* MOLECULAR DIAGNOSIS SEGMENT: Total bilirubin =< 2 x ULN (unless has Gilbert's disease) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* MOLECULAR DIAGNOSIS SEGMENT: Aspartate aminotransferase (AST)=< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* MOLECULAR DIAGNOSIS SEGMENT: Alanine aminotransferase (ALT) =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* MOLECULAR DIAGNOSIS SEGMENT: Creatinine clearance of >= 50 mL/min per 24-hour urine test or the Cockcroft-Gault formula (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* MOLECULAR DIAGNOSIS SEGMENT: If not receiving anticoagulants: international normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* MOLECULAR DIAGNOSIS SEGMENT: If not receiving anticoagulants: activated partial thromboplastin Time (aPTT) =<1.5 x ULN. If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* MOLECULAR DIAGNOSIS SEGMENT: Left ventricular ejection fraction (LVEF) >= 45% (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)

  * Note: Echocardiogram to be performed within 28 days prior to day 1 of protocol therapy
* MOLECULAR DIAGNOSIS SEGMENT: Corrected QT (QTc) =< 470 milliseconds (ms) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)

  * Note: Electrocardiogram (ECG) to be performed within 14 days prior to day 1 of protocol therapy
* MOLECULAR DIAGNOSIS SEGMENT: Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* MOLECULAR DIAGNOSIS SEGMENT: Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity from 4 weeks prior to first dose of treatment throughout the study treatment period and 1 month (females) or 1 month (males) from the last dose of study drug

  * Childbearing potential is defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* CHAPTER 1: Documented informed consent of the participant and/or legally authorized representative
* CHAPTER 1: Age: >= 18 years on the day of signing informed consent
* CHAPTER 1: ECOG =< 2
* CHAPTER 1: Patients with histologically confirmed AML, according to WHO criteria, with relapsed disease after alloHCT

  * Patients with non-central nervous system (CNS) extramedullary disease may be included if they also have marrow disease
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
* CHAPTER 1: Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 of prior anti-cancer therapy
* CHAPTER 1: White blood cell count less than 25 x 10^9 /L prior to initiation of venetoclax. Cytoreduction with hydroxyurea prior to treatment and/or up to 1 week after start of this treatment arm may be required (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 1: Total bilirubin =< 2 x ULN (unless has Gilbert's disease) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 1: AST =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 1: ALT =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 1: Creatinine clearance of >= 50 mL/min per 24-hour urine test or the Cockcroft-Gault formula (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 1: If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 1: If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 1: QTc =< 470 milliseconds (ms) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)

  * Note: ECG to be performed within 14 days prior to day 1 of protocol therapy
* CHAPTER 1: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* CHAPTER 1: Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity from 4 weeks prior to first dose of treatment throughout the study treatment period and 6 months (females) or 3 months (males) from the last dose of study drug

  * Childbearing potential is defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* CHAPTER 2: Documented informed consent of the participant and/or legally authorized representative
* CHAPTER 2: Age: >= 18 years on the day of signing informed consent
* CHAPTER 2: ECOG =< 2
* CHAPTER 2: Patients with histologically confirmed AML, according to WHO criteria, with relapsed disease after alloHCT

  * Patients with non-central nervous system (CNS) extramedullary disease may be included if they also have marrow disease
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
* CHAPTER 2: Patients with a confirmed susceptible FLT3 mutation (m) (internal tandem duplications (ITD), tyrosine kinase domain (TKD) mutations D835 or I836), or AXL variant expression
* CHAPTER 2: Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 of prior anti-cancer therapy
* CHAPTER 2: Total bilirubin =< 2 x ULN (unless has Gilbert's disease) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 2: AST =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 2: ALT =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 2: Creatinine clearance of >= 50 mL/min per 24-hour urine test or the Cockcroft-Gault formula (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 2: If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 2: If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 2: QTc =< 470 milliseconds (ms) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)

  * Note: ECG to be performed within 14 days prior to day 1 of protocol therapy
* CHAPTER 2: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* CHAPTER 2: Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity from 4 weeks prior to first dose of treatment throughout the study treatment period and 6 months (females) or 4 months (males) from the last dose of study drug

  * Childbearing potential is defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* CHAPTER 3: Documented informed consent of the participant and/or legally authorized representative
* CHAPTER 3: Age: >= 18 years on the day of signing informed consent
* CHAPTER 3: ECOG =< 2
* CHAPTER 3: Patients with histologically confirmed AML, according to WHO criteria, with relapsed disease after alloHCT

  * Patients with non-central nervous system (CNS) extramedullary disease may be included if they also have marrow disease
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
* CHAPTER 3: Patients with a confirmed susceptible BCR-ABL1 gene fusion
* CHAPTER 3: Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 of prior anti-cancer therapy
* CHAPTER 3: Total bilirubin =< 2 x ULN (unless has Gilbert's disease) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 3: AST =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 3: Creatinine clearance of >= 50 mL/min per 24-hour urine test or the Cockcroft-Gault formula (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 3: If not receiving anticoagulants: international normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 3: If not receiving anticoagulants: activated partial thromboplastin Time (aPTT) =<1.5 x ULN. If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 3: Left ventricular ejection fraction (LVEF) >= 45%

  * Note: Echocardiogram to be performed within 60 days prior to day 1 of protocol therapy
* CHAPTER 3: QTc =< 470 milliseconds (ms) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)

  * Note: ECG to be performed within 14 days prior to day 1 of protocol therapy
* CHAPTER 3: Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 3: Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity from 4 weeks prior to first dose of treatment throughout the study treatment period and 1 month (females) and 1 month (males) from the last dose of study drug

  * Childbearing potential is defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* CHAPTER 4: Documented informed consent of the participant and/or legally authorized representative
* CHAPTER 4: Age: >= 18 years on the day of signing informed consent
* CHAPTER 4: ECOG =< 2
* CHAPTER 4: Patients with histologically confirmed AML, according to WHO criteria, with relapsed disease after alloHCT

  * Patients with non-central nervous system (CNS) extramedullary disease may be included if they also have marrow disease
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
* CHAPTER 4: Patients with a confirmed susceptible IDH1 mutation (R132)
* CHAPTER 4: Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 of prior anti-cancer therapy
* CHAPTER 4: Total bilirubin =< 2 x ULN (unless has Gilbert's disease) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 4: AST =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 4: ALT =< 2 x ULN (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 4: Creatinine clearance of >= 50 mL/min per 24-hour urine test or the Cockcroft-Gault formula (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated in the study calendar)
* CHAPTER 4: If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (to be performed within 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-25 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Ability to obtain a molecular diagnosis (Molecular Diagnosis Segment) | From study enrollment to return of Molecular Diagnosis Report, assessed up to 30 days
  Outcome will be dichotomized based on return in =< 10 calendar days (Yes/No). Assessed by the proportion of successful participants.
Ability to make a treatment arm assignment by the Treatment Assignment Committee (TAC) (Molecular Diagnosis Segment) | From enrollment to treatment arm assignment by the TAC, assessed up to 30 days
  Outcome will be dichotomized based on return in =< 14 calendar days (Yes/No). Assessed by the proportion of participants who receive treatment assignment from TAC.
Incidence of adverse events (Treatment Segment) | Up to 30 days
  Toxicity will be graded according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Safety will be based on the assessment of dose limiting toxicity during cycle 1 and cycle 2. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Proportion of patients with successful sequencing (Molecular Diagnosis Segment) | Up to 30 days
  Successful sequencing is defined as passing quality control, and will be determined by City of Hope pathology among those with less than 20% blasts in the marrow aspirate.
Proportion of patients with successful treatment arm registration (Molecular Diagnosis Segment) | Up to 30 days
  Successful placement defined as the enrollment of a participant into one of the treatment arms.
Incidence of adverse events (Molecular Diagnosis Segment) | Up to 30 days
  Toxicity will be graded according to the NCI-CTCAE version 5.0. Safety will be based on the assessment of unacceptable toxicity during glasdegib monotherapy. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Overall response (Treatment Segment) | Up to the date of the first of 2 successive bone marrows showing said response, assessed up to 30 days
  Response will be based on Dohner et al., 2017 criteria. Response dates recorded will be the date of the first of 2 successive bone marrows showing said response. For this trial, will assess the complete remission rate calculated as the percent of evaluable patients that have confirmed complete response (CR) or incomplete blood count recovery (CRi). 95% Clopper Pearson binomial confidence interval will be calculated. Response rates will also be explored based on number/type of prior therapy(ies).
Duration of remission (Treatment Segment) | Time from the first of two consecutive bone marrow aspirates showing CR or CRi until such time as the bone marrow or peripheral blood mononuclear cells shows signs of relapse, assessed up to 30 days

OTHER OUTCOMES:
Change in leukemia stem cell (LSC) burden (Treatment Segment) | Baseline up to post-treatment (2 cycles) (each cycle = 28 days)
  Measured by limiting dilution and engraftment into non-obese diabetic severe combined immunodeficiency gamma severely immunocompromised mice. Graphical statistics will be used. To assess the association between the LSC reduction and the response to the treatment, the median change from baseline to post-treatment (2 cycles) in engraftment levels of secondary mice recipients (n=12 mice/patient, 6 females and 6 males) will be compared by two-sample t test between response and non-response patient groups as LSC donors, across all treatment arms. The effect of treatment on the target genes will be assessed for each arm by linear mixed models (pre- versus multiple post-treatment time points) as well.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Meidcal Center, Duarte, California, United States